CLINICAL TRIAL: NCT06098885
Title: The Effect of Different Treatment Modalities of Class II Malocclusion on Upper Third Molars: A Retrospective Longitudinal Study
Brief Title: The Effect of Different Treatment Modalities of Class II Malocclusion on Upper Third Molars.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Aboalnaga, principal investigator, Cairo University
Other Study IDs: CEBD-CU-2021-9-7
Record Dates: First submitted 2021-09-08; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Third Molar Impaction
Keywords: distalization; premolar extraction; upper third molar; impaction of third molar

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- extraction treatment: patients treated with bilateral upper first premolar extraction orthodontic treatment with moderate anchorage.
  Interventions: Other: extraction orthodontic treatment
- distalization treatment: patients treated by distalization orthodontic treatment.

INTERVENTIONS:
Other: extraction orthodontic treatment — bilateral upper first premolar extraction orthodontic treatment with moderate anchorage.
  Groups: extraction treatment

SUMMARY:
What is the effect of the different treatment modalities (distalization versus upper premolar extraction) of class II malocclusion on the position, inclination and incidence of impaction of the upper third molars?

DETAILED DESCRIPTION:
What is the effect of the different treatment modalities (distalization versus upper premolar extraction) of class II malocclusion on the position, inclination and incidence of impaction of the upper third molars? Pico P: Adolescent patients with class II malocclusion having bilateral developing upper third molars.

I: bilateral upper first premolar extraction orthodontic treatment with moderate anchorage.

C: distalization orthodontic treatment. O: Primary: angulation of the maxillary third molars.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent males and females (16 -18 years) with Bilaterally developing maxillary third molars. Not more than two thirds of the root development of the third molars had taken place.
* Class II malocclusion cases that were treated by 1) maxillary premolar extraction with a moderate anchorage requirement and achieved full unit class II molar relationship or 2) Distalization treatment plan and class I molar relationship was achieved.
* Patients with high-quality pre- and post-treatment radiographs.
* Normal or increased vertical dimension.

Exclusion Criteria:

* Maxillary Premolar extraction cases requiring maximum anchorage preparation.
* Low vertical dimension.
* Patients without dentofacial deformities, severe facial asymmetries, microdontia or hypodontia.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: • Egyptian Adolescent males and females (16 -18 years)
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-06-04 (Actual)

PRIMARY OUTCOMES:
The angulation of the maxillary third molars. | up to 24 weeks.
  the angle between the long axis of the third molar and the palatal plane

SECONDARY OUTCOMES:
The vertical position of the third molars | up to 24 weeks
  the vertical position of the third molar relative to the second molar measured using Archer classification tool. (qualitative measure)
The mineralization status of the third molars | up to 24 weeks
  the amount of calcified tissues of the third molar measured using Demirjian classification method

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Aboalnaga, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided